CLINICAL TRIAL: NCT03287167
Title: A Prospective, Double -Blind ,Multi-center,Randomized Controled Trial of Comparison One vs Six Months of Dual Antiplatelet Therapy After Implanted Sirolimus- Eluting Stent With Abluminal Grooves Containing A Biodegradable Polymer (FirehawkTM Stent ) in High Bleeding Risk Patients With Coronary Artery Disease
Brief Title: Comparison One vs Six Months of Dual Antiplatelet Therapy After Implanted Firehawk TM Stent in High Bleeding Risk Patients With Coronary Artery Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TARGET SAFE
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Coronary Disease; Drug Eluting Stent; Percutaneous Coronary Intervention; Dual Antiplatelet Therapy
MeSH Terms: conditions — Coronary Disease | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 month DAPT intervention (Experimental): After implantation of Firehawk coronary stents, 860 subjects in intervention group will be given dual anti-platelet therapy (DAPT) including aspirin and clopidogrel for 1 month， then will be given aspirin and placebo for next 5 months.
  Interventions: Drug: 1 month DAPT
- 6 months DAPT intervention (Active Comparator): After implantation of Firehawk coronary stents, 860 subjects in control group will be given dual anti-platelet therapy (DAPT) including aspirin and clopidogrel for 6 months.
  Interventions: Drug: 6 months DAPT

INTERVENTIONS:
Drug: 1 month DAPT — Subjects will continue DAPT with clopidogrel and Aspirin (ASA) up to 1 month, after which patients will be given ASA and placebo in next 5 months and then continue on monotherapy with ASA only, unless contraindications for ASA emerge.
  Arms: 1 month DAPT intervention
Drug: 6 months DAPT — Subjects will continue DAPT with clopidogrel and Aspirin (ASA) up to 6 months, after which patients will continue on monotherapy with ASA only, unless contraindications for ASA emerge.
  Arms: 6 months DAPT intervention

SUMMARY:
This study is to assess the clinical non-inferiority of 1 month (short-term) vs 6 months (long-term) of dual anti-platelet therapy in patients undergoing percutaneous intervention implanted sirolimus -eluting stent with abluminal grooves containing a biodegradable polymer in High Bleeding Risk patients with coronary artery disease.

DETAILED DESCRIPTION:
This is a prospective, double -blind,multi-center,randomized controlled trial. Approximately 1,720 subjects in high bleeding risk with coronary artery disease will be enrolled in no more than 40 research centers in China. All participants met the inclusion criteria will be 1:1 randomized to 1 month or 6months of DAPT after implanting Firehawk™ coronary stent. Clinical follow-up will be carried out at 30 days, 6 months, 12 months, 2 years after index procedure.The primary study endpoint is Net Adverse Clinical and Cerebral Events (NACCE), a composite of all-cause death, myocardial infarction (MI), cerebral vascular accident (CVA) and major bleeding ([BARC] definition) at 12 months. Subjects that complete of 12 months follow-up will be regarded as having completed the primary endpoint. The secondary study endpoints contain cost-effectiveness at 12 months, ARC defined stent thrombosis (ST) ; NACCE ;major adverse cardiovascular events (MACE),major adverse cardiovascular and cerebral events (MACCE),target lesion revascularization (TLR),target vessel failure(TVF) , major bleeding at 30 days,6,12 and 24 months of follow-up.

ELIGIBILITY:
General Inclusion Criteria:

* Age ≥ 18 years;
* Subjects (or legal guardians) understand the testing requirements and procedures, and provide written informed consent;
* Subjects could undergo percutaneous coronary intervention (PCI);
* Subjects have symptomatic coronary artery disease or have confirmed asymptomatic ischemia;
* Subjects are eligible candidates for coronary artery bypass graft surgery (CABG);
* Left ventricular ejection fraction (LVEF) within 60 days ≥ 30%;
* Subjects were willing to accept the trial plan calls for all subsequent evaluations;
* Subjects can endure 6 months dual anti-platelet therapy, and met one or more criteria as the following:

  1.Age ≥ 75years; 2.Subjects with hemoglobin<10g/dL, or subjects received transfusion therapy 4 weeks ago; 3.Subjects with renal insufficiency (eGFR < 60 ml / min); 4. Subjects with HAS-BLED score ≥3.0; 5.Femal patients with acute cononary syndrome; 6.BMI < 18.5 Kg/M2; 7.Subjects with congestive heart failure and with LVEF30%-50%; 8.Subjects had a history of hospitalization due to bleeding; 9.Subjects with thrombocytopenia (platelet < 100,000 / mm3); 10.Subjects had a histroy of intracranial hemorrhage; 11.Subjects had a histroy of intracranial ischemia stroke in 6 months; 12.Subjects plan to receive non-steroidal anti-inflammatory or steroid treatment for more than 30 days after the baseline PCI; 14.Subjects were expected to receive additional treatment after PCI and cannot undergo long-term DAPT therapy; 15.Subjects had a history of stomach ulcers or active ulcers.

Angiographic Inclusion Criteria

* Target lesions must be new and have a visually estimated reference diameter ≥2.25 mm and ≤4.0 mm in autologous coronary artery;
* Target lesions must be moderate-severe calcification;
* No limitations in target lesion length and number, and the number of implanted stents is less than 4;
* ALL target lesion must be able to successfully expand and implant Firehawk™ stent.

Clinical Exclusion Criteria:

* Subjects recently suffer from MI (within 4 week) and ECG changes/clinical symptoms consistent with AMI, or accompanied with increased cardiac biomarkers (CK-MB, CK, TNT or TNI) and at least one of the following :

  1. CK-MB> 3ULN, regardless of the value of total CK;
  2. If CK-MB or CK was not detected, but cTN> 1ULN, and at least one of the following:

     1. Ischemic symptoms and ECG changes of new ischemia;
     2. Development of pathologic Q waves in the ECG;
     3. Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.
* Subject had Re-MI before randomized;
* Subject with hemodynamic instability (Killip class IV);
* Subjects were detected ventricular aneurysm greater than 3.0*2.0cm or intraventricular thrombosis by cardiac ultrasonography in 30 days;
* Subjects with Life-threatening arrhythmias;
* Subjects were expected to receive oral anticoagulation therapy after the baseline PCI;
* Subjects cannot endure dual anti-platelet therapy for 1 month;
* Subjects with mechanical complications after myocardial infarction;
* Subjects had an organ transplant or are waiting for an organ transplant;
* Subjects are receiving chemotherapy or will receive a chemotherapy within 30 days after PCI;
* Subjects with abnormal counts of white blood cell (WBC);
* Subjects with verified or suspected acute liver disease, including lab results of acute liver disease;
* Subjects had permanent neurological diseases in the past 6 months;
* Subjects had any PCI (such as balloon angioplasty, stent, cutting balloon) treatment in target vessels within 12 months prior to baseline;
* Non-target vessel had been implanted non-research stent 5 months ago before the baselin PCI.
* Subjects plan to undergo PCI or CABG within 1 year after the baseline PCI;
* Subjects have any coronary endovascular brachytherapy treatment previously;
* Subjects associated with drugs allergy (such as sirolimus, or structure-related compounds fluorinated polymers, thiophenepyridine or aspirin);
* Subjects are suffering from other serious illness (such as cancer, congestive heart failure), which may cause drop in life expectancy to less than 12 months;
* Subjects are currently abusing drugs (such as alcohol, cocaine, heroin, etc);
* Subject plan to undergo any operations that may lead to confuse with the programme;
* Subjects were participating in another study of drug or medical device which did not meet its primary endpoint;
* Subjects plan to pregnant within 12 months after baseline;
* Subjects are pregnant or breastfeeding women.

Angiographic Exclusion Criteria (visual estimate):

* Target lesions with the following criteria: left main, saphenous vein grafts or arterial grafts, via saphenous vein grafts or arterial graft, more than 4 stents have been implanted and in-stent sestenosis;
* Subjects with unprotected left main coronary artery disease (diameter stenosis >50%);
* Subjects have a protected left main coronary artery disease (diameter stenosis> 50% and left coronary artery bypass surgery), as well as target lesions located in the LAD and LCX;
* Subjects with other lesions of clinical significance, may be need intervention within 12 months after baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1720 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Net Adverse Clinical and Cerebral Events (NACCE) | At 12 months after index procedure
  A composite of all-cause death, MI, cerebral vascular accident (CVA) and major bleeding at 18 months

SECONDARY OUTCOMES:
Target Vessel Revascularization (TVR) | In hospital and at 30 days,6, 12 and 24 months after index procedure
Target lesion Revascularization (TLR) | In hospital and at 30 days,6, 12 and 24 months after index procedure
Target Vessel Failure (TVF) | In hospital and at 30 days,6, 12 and 24 months after index procedure
Target Lesion Failure (TLF) | In hospital and at 30 days,6, 12 and 24 months after index procedure
Stent Thrombosis (per ARC definition) | In hospital and at 30 days,6, 12 and 24 months after index procedure
  the definite and probable stent thrombosis
Major Adverse Cardiac and Cerebral Events(MACCE) | In hospital and at 30 days,6, 12 and 24 months after index procedure
Net Adverse Clinical and Cerebral Events (NACCE) | In hospital and at 30 days,6, 12 and 24 months after index procedure
Myocardial Infarction (MI,including Q-wave MI and non Q-wave MI) | In hospital and at 30 days,6, 12 and 24 months after index procedure
Death (All cause, Cardiac, Non-cardiac) | In hospital and at 30 days,6, 12 and 24 months after index procedure
Cardiac Death | In hospital and at 30 days,6, 12 and 24 months after index procedure
Non-Cardiac Death | In hospital and at 30 days,6, 12 and 24 months after index procedure
Major Bleeding | In hospital and at 30 days,6, 12 and 24 months after index procedure
  [BARC] definition

OTHER OUTCOMES:
Cost-Effectiveness Ratio (CER) | At 12 months after index procedure
  CER = [total medical care costs of anti-platelet therapy] / [number of participants without net adverse clinical and cerebral events (NACCE)]

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — The General Hospital of Shenyang Military
Locations (1):
- The General Hospital of Shenyang Military, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices) will be shared. Additionally, study protocol will be available. The data will become available for the beginning 3 months and ending 5 years following article publication. The access criteria are as follow:
  (With) Researchers who provide a methodologically sound proposal. (For the analysis) to achieve aims in the approved proposal. (Requisite mechanism) Proposals should be directed to mzheng@microport.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).
  If the data sharing plan changes after registration, this should be reflected in the statement submitted and published with the manuscript, and updated in the registry record.
Supporting Information: Study Protocol
Time Frame: Beginning 1 months and ending 5 years following article publication
Access Criteria: (With) Researchers who provide a methodologically sound proposal. (For the analysis) to achieve aims in the approved proposal. (Requisite mechanism) Proposals should be directed to mzheng@microport.com. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link to be included).

REFERENCES:
- [Derived] Lee SH, Kim J, Lefieux A, Molony D, Shin D, Hwang D, Choi KH, Chang HS, Jeon KH, Lee HJ, Jang HJ, Kim HK, Ha SJ, Park TK, Yang JH, Song YB, Hahn JY, Choi SH, Doh JH, Shin ES, Nam CW, Koo BK, Gwon HC, Lee JM. Clinical and Prognostic Impact From Objective Analysis of Post-Angioplasty Fractional Flow Reserve Pullback. JACC Cardiovasc Interv. 2021 Sep 13;14(17):1888-1900. doi: 10.1016/j.jcin.2021.07.014. PMID 34503739
- [Derived] Capodanno D. Another Coronary Stent for Patients at High Bleeding Risk. JACC Cardiovasc Interv. 2021 Sep 13;14(17):1884-1887. doi: 10.1016/j.jcin.2021.07.028. No abstract available. PMID 34503738